CLINICAL TRIAL: NCT00837967
Title: A Comparison of Tolerability of 10 Inhalations of Symbicort® Turbuhaler® 160/4.5 μg and 10 Inhalations of Terbutaline Turbuhaler® 0.4 mg on Top of Symbicort® Turbuhaler® 160/4.5 μg 1 Inhalation Bid, Randomized, Double-blind, Cross Over, Phase III Study in Japanese Adults Asthma Patients
Brief Title: Study to Investigate the Safety and Efficacy of High Dose of Symbicort® SMART in Japanese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D589LC00003
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
Keywords: Asthma; Symbicort Turbuhaler
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Symbicort, then Terbutaline (Experimental): Symbicort Turbuhaler 160/4.5μg for 3 days First , then Terbutaline Turbuhaler 0.4 mg for 3 days
  Interventions: Drug: Symbicort Turbuhaler; Drug: Terbutaline Turbuhaler
- First Turbuhaler, then Symbicort (Experimental): Terbutaline Turbuhaler 0.4 mg for 3 days First, then Symbicort Turbuhaler 160/4.5μg for 3 days,
  Interventions: Drug: Symbicort Turbuhaler; Drug: Terbutaline Turbuhaler

INTERVENTIONS:
Drug: Symbicort Turbuhaler — 160/4.5μg for 3 days
Drug: Terbutaline Turbuhaler — 0.4 mg for 3 days

SUMMARY:
The primary objective of the study is to compare the tolerability of Symbicort® Turbuhaler® 160/4.5 μg 10 inhalations with terbutaline Turbuhaler® 0.4 mg 10 inhalations for 3 days on top of Symbicort® Turbuhaler® 160/4.5 μg 1 inhalation twice a day (bid) in adult asthma patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* A minimum of 6 months documented history of asthma according to the JGL2006/GINA2006 definition
* FEV1> 70% of predicted normal value pre-bronchodilator

Exclusion Criteria:

* Having a known or suspected allergy to study therapy (active drugs or additive)
* Having a known clinical history of hypertension, relevant arrhythmias or other heart disease, eg, ischemic heart disease, cardiomyopathy, valvular heart disease, or heart failure
* Having been treated with oral, parenteral or rectal glucocorticoids within 4 weeks, or with depot parenteral glucocorticoids within 3 months
* Respiratory infection significantly affecting the asthma, as judged by the investigator within 4 weeks

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Andersson, MD, Study Director — AstraZeneca R&D Lund
Locations (2):
- Japan (2):
  - Research Site, Ibaraki
  - Research Site, Tokyo

REFERENCES:
- [Derived] Saito T, Hasunuma T. Safety and tolerability of high-dose budesonide/formoterol via Turbuhaler(R) in Japanese patients with asthma: a randomized, double-blind, crossover, active comparator-controlled, phase III study. Clin Drug Investig. 2012 Jan 1;32(1):51-61. doi: 10.2165/11595440-000000000-00000. PMID 22024920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from 2 hospitals in Japan between January 2009 and July 2009. 28 patients enrolled; 25 patients randomized, 3 patients were not randomized (1 due to incorrect enrollment and 2 due to adverse event)
Groups:
- Symbicort First, Then Terbutaline: Symbicort Turbuhaler 160/4.5μg for 3 days First , then Terbutaline Turbuhaler 0.4 mg for 3 days
- Terbutaline First, Then Symbicort: Terbutaline Turbuhaler 0.4 mg for 3 days First, then Symbicort Turbuhaler 160/4.5μg for 3 days,
Period: First Intervention
Arm/Group | Symbicort First, Then Terbutaline | Terbutaline First, Then Symbicort
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: Washout Period of 7 - 14 Days
Arm/Group | Symbicort First, Then Terbutaline | Terbutaline First, Then Symbicort
Started | 13 | 12
Completed | 11 | 12
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Second Intervention
Arm/Group | Symbicort First, Then Terbutaline | Terbutaline First, Then Symbicort
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 44.3 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Total number of adverse events
Time Frame: 3 days
Measure: Number; unit: adverse events
Groups:
- Symbicort: Symbicort Turbuhaler 160/4.5μg
- Terbutaline: Terbutaline Turbuhaler 0.4 mg
Arm/Group | Symbicort | Terbutaline
Number analyzed (Participants) | 25 | 23
adverse events | 14 | 24

2. Primary Outcome: Serum Potassium - Average Concentration From Trapezoidal Area Under the Curve (AUC)
Description: The mean AUC value was calculated as AUC (calculated using the trapezoidal method) divided by the length of the sampling period.
Time Frame: up to 740 min after start dosing for each treatment day
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Symbicort | Terbutaline
Number analyzed (Participants) | 25 | 23
mEq/L | 4.01 (0.25) | 3.88 (0.26)

3. Primary Outcome: Blood Glucose - Average Concentration From Trapezoidal Area Under the Curve (AUC)
Description: as for outcome 2
Time Frame: up to 140 min after start dosing for each treatment day
Measure: Mean (Standard Deviation); unit: mg/dLiters
Arm/Group | Symbicort | Terbutaline
Number analyzed (Participants) | 25 | 23
mg/dLiters | 121.1 (20.3) | 129.5 (22.0)

4. Primary Outcome: Electrocardiogram (ECG)- Average Trapezoidal Area Under the Curve (AUC)
Description: The mean AUC of QTcF (ECG interval measured from the beginning of the Q wave to the end of the T wave, corrected for heart rate using Fridericia's formula)was calculated as AUC (calculated using the trapezoidal method) divided by the length of the sampling period.
Time Frame: up to 740 min after start dosing for each treatment day
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Symbicort | Terbutaline
Number analyzed (Participants) | 25 | 23
ms | 411.71 (15.07) | 414.33 (14.04)

5. Primary Outcome: Vital Sign (Blood Pressure)- Average Trapezoidal Area Under the Curve (AUC)
Description: as for outcome 2
Time Frame: up to 740 min after start dosing for each treatment day
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Symbicort | Terbutaline
Number analyzed (Participants) | 25 | 23
mmHg | 115.3 (6.3) | 114.9 (8.0)

6. Primary Outcome: Vital Sign (Pulse Rate)- Average Trapezoidal Area Under the Curve (AUC)
Description: as for outcome 2
Time Frame: up to 740 min after start dosing for each treatment day
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Symbicort | Terbutaline
Number analyzed (Participants) | 25 | 23
beats/min | 70.0 (6.6) | 74.1 (7.5)

ADVERSE EVENTS:
Description: Of 25 patients in safety analysis set, 2 patients did not receive terbutaline due to adverse events lead to discontinuation. Therefore, data from 25 patients for Symbicort and 23 patients for terbutaline were used for the safety evaluation.
Groups:
- Symbicort: Symbicort Turbuhaler 160/4.5μg for 3 days
- Terbutaline: Terbutaline Turbuhaler 0.4 mg for 3 days
Arm/Group | Symbicort | Terbutaline
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 7/25 | 15/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort (N=25) | Terbutaline (N=23)
Nasopharyngitis (Infections and infestations) | 2 | 2
Tremor (Nervous system disorders) | 3 | 4
Palpitations (Cardiac disorders) | 1 | 3
Tachycardia (Cardiac disorders) | 1 | 3
Blood Pressure Decreased (Investigations) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No